CLINICAL TRIAL: NCT03265418
Title: BioXmark Liquid Fiducials to Enable Radiotherapy Tumor Boosting in Rectal Cancer, a Feasibility Trial
Brief Title: BioXmark, Rectal Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W 16 09 00091
Record Dates: First submitted 2017-04-26; First posted 2017-08-29 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — X-Rays; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BioXmark liquid fiducial markers (Experimental): Placement of 4 BioXmark liquid fiducial markers, standard treatment (chemo-radiotherapy followed by surgery or wait-and-see) with extra imaging to evaluate the behaviour of the markers before, during and after the radiotherapy
  Interventions: Device: BioXmark liquid fiducial markers; Other: Imaging; Procedure: surgery or wait-and-see

INTERVENTIONS:
Device: BioXmark liquid fiducial markers — Before the start of the treatment planning during an extra sigmoidoscopy after enema preparation, 4 liquid marker spots will be placed 1 cm from the tumor; two in the in the cranial and two in the caudal direction of the tumor (4 markers in total per patient).
Other: Imaging — As part of standard patient set-up directly before each radiotherapy treatment, kV cone-beam CTs will be acquired. Treatment positioning will be based on the regular clinical decision protocols for treatment of rectal cancer and not on the markers. During treatment potential fiducial movement will be assessed using an externally positioned ultra-sound probe, positioned against the abdominal or perineal skin of the patients depending on de position of the tumor/fiducials in the rectum. For patients in this study 2 orthogonal kV images will be made immediately after each radiation using the electronic portal imaging (EPI) device.
  As part of standard clinical practice an MR of the rectum will be made for response evaluation 6-8 weeks after the end of neo-adjuvant chemo-radiotherapy.
Procedure: surgery or wait-and-see — As part of standard clinical practice patients whose tumor has not responded completely will be operated on 8-12 weeks after the end of neoadjuvant chemo-radiotherapy. Patients with a complete response will be follow-upped according to the "wait-and-see" protocol.

SUMMARY:
To test the feasibility and accuracy of BioXmark fiducial markers for image guided radiotherapy (IGRT) based rectal tumor boosting in 20 patients referred for long course chemo-radiotherapy of the locally advanced rectal cancer.

DETAILED DESCRIPTION:
This study is a prospective non-randomized open label trial.

A total of 20 patients who will undergo neo-adjuvant chemo-radiotherapy for rectal cancer will be included in this study upon informed consent.

During an extra sigmoidoscopy after enema preparation, 4 liquid marker spots will be placed 1 cm from the tumor; two in the in the cranial and two in the caudal direction of the tumor (4 markers in total per patient).

Participants will undergo standard treatment for their rectal cancer.

As part of standard patient set-up directly before each radiotherapy treatment, kilovoltage (KV) cone-beam computed tomography (CBCT) will be acquired. Treatment positioning will be based on the regular clinical decision protocols for treatment of rectal cancer and not on the markers. During treatment potential fiducial movement will be assessed using an externally positioned ultra-sound probe (this probe will be positioned against the abdominal or perineal skin of the patients depending on de position of the tumor/fiducials in the rectum). Moreover, for patients in this study 2 orthogonal kV images will be made immediately after each radiation using the electronic portal imaging (EPI) device.

As part of standard clinical practice an Magnetic resonance imaging (MRI) of the rectum will be made for response evaluation 6-8 weeks after the end of neo-adjuvant chemo-radiotherapy.

As part of standard clinical practice patients whose tumor has not responded completely will be operated on 8-12 weeks after the end of neoadjuvant chemo-radiotherapy. Patients with a complete response will be follow-upped according to the "wait-and-see" protocol.

Cone-beam CT and MR images which are obtained as routine practice during treatment of the participants will be compared with images of 20 non-participating patients treated at our institute in the same period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological or cytological proven adenocarcinoma of the rectum, treated with long course external beam radiotherapy
* Age > 18 years
* Have given written informed consent before patient registration

Exclusion Criteria:

* Patients using anticoagulants: platelet aggregation inhibitors or coumarines
* Iodine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Positional stability of BioXmark liquid fiducial markers during the treatment course | will be determined through the course of radiotherapy, an average of 5 weeks
  Positional stability / potential marker migration will be assessed by calculating marker pair distances.

SECONDARY OUTCOMES:
Visibility/visual stability of BioXmark liquid fiducial markers during the treatment course | will be determined for the time interval between placement and the post-treatment MRI, an average of 12 weeks
  Visual stability will be evaluated by scoring visibility of the markers on CT, CBCT, EPI and MRI (T1, T2 and diffusion weighted images) by 2 independent observers using a subjective scoring system: 0 = not visible, 1 = barely visible, 2 = clearly visible.
Percentage of markers lost from injection to CT acquisition for RT planning | will be determined for the time interval between placement and pretreatment radiotherapy planning CT, an average of 1 week
  (1 - number of markers visible on the last CBCT (cone-beam computed tomography) during treatment / number of visible markers at pCT) * 100
Percentage of markers lost from injection to CT acquisition for RT planning | will be determined for the time intervals through the course of radiotherapy, an average of 5 weeks
  (1 - number of markers visible on the last CBCT (cone-beam computed tomography) during treatment / number of visible markers at pCT) * 100
Adverse events (AE) potentially associated with BioXmark | until rectal surgery, on average 11 weeks, or in case of omission of surgery, until 3 months after marker placement.
  The safety of bioXmark liquid fiducials placement will be assessed by recording Adverse events (AE) potentially associated with BioXmark until rectal surgery, on average 11 weeks, or in case of omission of surgery, until 3 months after marker placement.
Inter-observer variation in gross tumor volume (GTV) localization with and without markers | through the course of radiotherapy, an average of 5 weeks
  The concordance index (CI) of gross tumor volume (GTV) localization between observers on kV CBCT will be determined. The CI is the ratio of the intersection and the union of the two volumes.
Effect of BioXmark liquid fiducial markers on post-treatment MRI images | at the moment of the post-treatment MRI, on average 6-8 weeks after chemo-radiation
  Potential BioXmark induced artefacts will be scored by 2 independent observers using a subjective scoring system:
Potential BioXmark induced alterations in the surgical specimen | on average 10-12 weeks after chemo-radiation
  The surgical specimens will be evaluated for signs of marker-induced alterations.
  Potential BioXmark induced alteration in the surgical specimen will be scored by 2 independent observers using a subjective scoring system.In case the markers can't be located in the surgical specimen standard clinical evaluation of the specimen will take place. If the marker got lost during tissue processing potential inflammation/perforation will be scored as follows:A) 0 = no signs of extra inflammatory changes possibly related to the fiducials, 1 = limited extra inflammatory changes possibly related to the fiducials, 2 = severe extra inflammatory changes possibly related to the fiducials; B) 0 = no perforation of the rectal possibly related to fiducials, 1 = perforation of the rectal possibly related to the fiducials

CONTACTS AND LOCATIONS:
Overall Officials: Maaike Berbée, MD,PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO Clinic, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No